CLINICAL TRIAL: NCT05332977
Title: Clinical Performance, Patient and Operator Reported Outcome Measures of Axially Placed and Tilted Implants Used for Fixed Rehabilitation of the Edentulous Maxilla.
Brief Title: Clinical Study Investigating the Efficiency and Complications Related to Two Different Procedures Used for the Preparation of Dentures Applied in Patients With Edentulous
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: ITI Foundation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAD-CAM vs DC
Record Dates: First submitted 2022-01-28; First posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Edentulous Maxilla
Keywords: CAD-CAM integrating digital workflow

STUDY DESIGN:
Intervention Model Description: The edentulous patients recruited in the study will be randomized into the following two groups:
  * Placement of tilted implants in the distal most position (group-Til) with straight implants in the anterior region
  * Placement of axial implants in the distal most position (group-Axl) with straight implants in the anterior region
  Subjects from the above groups will be further divided into following two sub-groups:
  * Immediate loading using denture conversion prosthesis (group DC)
  * Immediate loading using milled PMMA prosthesis (group CAD-CAM)
Who Masked: Participant
Masking Description: As the placement of implants and the type of implant is clearly distinguishable and require different handling, blinding of the prosthodontist is not feasible.
  Patients are blinded to the type of implant received and to the type of procedure followed for the fabrication of the provisional prosthesis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAD-CAM fabricated provisional prothesis (Experimental): Insertion of CAD-CAM fabricated provisional prosthesis (CAD-CAM) on axially placed or titled implants for rehabilitation of atrophic maxilla
  Interventions: Device: CAD-CAM fabricated provisional prosthesis
- Insertion of denture conversion (DC) (Active Comparator): Insertion of denture conversion (DC) provisional prosthesis on axially placed or titled implants for rehabilitation of atrophic maxilla
  Interventions: Device: DC (denture conversion) provisional prosthesis

INTERVENTIONS:
Device: CAD-CAM fabricated provisional prosthesis — Insertion of CAD-CAM fabricated provisional prosthesis (CAD-CAM) on axially placed or titled implants for rehabilitation of atrophic maxilla
  Arms: CAD-CAM fabricated provisional prothesis
Device: DC (denture conversion) provisional prosthesis — Insertion of denture conversion (DC) provisional prosthesis on axially placed or titled implants for rehabilitation of atrophic maxilla
  Arms: Insertion of denture conversion (DC)

SUMMARY:
The principal aim of the study is to evaluate the prosthetic complications with CAD-CAM fabricated provisional prostheses and denture conversion prostheses after 3 months of function. Supported restorations are now a predictable treatment modality for the rehabilitation of complete and partially edentulous jaws.Immediate loading of the placed implants is performed for the rehabilitation of the edentulous arch to improve patients' function. This can be usually done by converting the existing denture base of the patient or by making a CAD- CAM milled provisional prosthesis integrating digital workflow. A laboratory fabricated denture base can be converted into a screw-retained provisional prosthesis post implant placement. This is known as conversion prosthesis. However, drawbacks of these prostheses include increased chairside time for the clinician leading to inconvenience for the patient and a potential for an error in prosthesis fabrication. With the introduction of CAD-CAM technology, it is now possible to fabricate a provisional restoration using digital workflows. This workflow would help the clinicians save a considerable amount of chairside time and obtain potentially stronger restorations better polished and without contamination of surgical field. Studies assessing the soft tissue response and patient-reported outcome measures between denture conversion and CAD- CAM fabricated provisionals are currently lacking in the literature.

DETAILED DESCRIPTION:
1. Study Intervention and Indication CAD-CAM fabricated provisional prostheses facilitate prosthesis delivery in immediate functional loading protocols. The prostheses are manufactured in the laboratory by milling high-density polymers based on a highly cross-linked polymethylmethacrylate (PMMA). The prostheses are known to have higher biocompatibility, superior esthetics and soft tissue response as compared to denture conversion prostheses.

   The indication is edentulism. CAD-CAM fabricated prostheses are implant supported prosthesis and are indicated for rehabilitation of edentulous arch.
2. Justification of Study Intervention With the introduction of CAD-CAM technology, it is now possible to fabricate a provisional restoration using digital workflows. This workflow would help the clinicians to save a considerable amount of chairside time and to obtain potentially stronger restorations better polished and without contamination of surgical field.
3. Risk / Benefits The participants will be exposed to only minor risks (loosening of prosthesis), as all procedures used in this study for rehabilitation of the patients have been used in dental clinics. The safety and risk profiles are well known. Patients will be locally anesthetized during the procedure of implant placement. Well-experienced dentists who are very familiar with the procedures and materials used will perform the surgeries. On the other hand, a significant gain of knowledge will be expected by the use of CAD-CAM fabricated and denture conversion provisional prostheses. This will open new insights in respect to rehabilitation of the patients undergoing full arch reconstructions. Consequently, this will open new therapeutical opportunities in order to provide the best and most adequate treatment strategy for future patients.

   It is ethically justifiable that the patients included in this study will receive the CAD-CAM fabricated provisional prosthesis as well as the denture conversion prosthesis as this represents todays standard and most often performed procedure.

   Anticipated adverse effects and residual risks encompass loosening of the prosthesis.
4. General Study Design and Justification of the design This study will be designed as monocenter prospective randomized, controlled, clinical trial with two parallel study groups and a follow-up duration of 5 years after insertion of the final prostheses.

   Treatment interventions and follow-up:

   The edentulous patients recruited in the study will be randomized into the following two groups:
   * Placement of tilted implants in the distal most position (group-Til) with straight implants in the anterior region
   * Placement of axial implants in the distal most position (group-Axl) with straight implants in the anterior region

   Subjects from the above groups will be further divided into following two sub-groups:
   * Immediate loading using denture conversion prosthesis (group DC)
   * Immediate loading using milled PMMA prosthesis (group CAD-CAM)
5. Methods of Minimising Bias As the implants are clearly distinguishable and require different handling, blinding of the surgeon is not feasible.

   The patients will be given questionnaires and they will be asked to answer them before the start of each visit in absence of the investigator or any study site team member.

   Additionally, the patients are informed about two different procedures for the fabrication of the provisional prosthesis; however, they are not told about the technical details and which fabrication workflow they have been allocated.

   The ease of insertion of the provisional prostheses will be evaluated by an evaluator other than the surgeon. This evaluator will be the same for both prostheses throughout the study.
6. Assignment to Study Group Axial or Tilted implants will be allocated randomly to the patients, so that an equal distribution (1:1) of patients to both treatment groups results. Similarly, patients will be randomly allocated to group DC and group CAD-CAM prosthesis. The randomization sequences will be generated by using a computer-generated list. The study manager or the statistician will generate the allocation sequences and will store them with restricted access. One randomization will be done by the eCRF after uploading the allocation list and the other randomization will be performed by opening sealed envelopes Whenever an investigator enrolls a patient for the study, a subject number (ordered number given by the system with a center identification code) will be assigned to the patient. Subject number will be recorded on the medical record folder of the patient. Subject identification Log will enable direct connection to patient identity. This list will be filed in a folder with limited access only for study members and will be kept on site.
7. Monitoring Institution Due to the minimal risk of the study (all treatments are performed according to the standard of care) no external monitoring is needed.

   The quality control will be performed by an internal study monitor of M.A. Rangoonwala College of Dental Sciences. If needed, remote monitoring will be performed by the study management team located in Zurich.
8. Statistical Methods

Hypothesis

The hypothesises of the present RCT are two-fold:

1. There will be no differences in the prosthetic complications of CAD-CAM fabricated provisionals and denture conversion prostheses (DC) when used as provisional prostheses.
2. There will be no difference in the survival rates between tilted and axially placed short implants in distal positions for the rehabilitation of the edentulous maxilla with fixed screw-retained prostheses.

Determination of Sample Size Sample size was determined using the percentage of prosthetic complications observed in previous clinical trials, using the formula, n = 2 (Zα+ Zβ)2 p(1-p) d2

where Zα is the z variate of alpha error i.e. a constant with value 1.96, Zβ is the z variate of beta error i.e. a constant with value 0.84, p is the proportion of events

Approximate estimates:

1. 80% power
2. Type I error to be 5%
3. Type II error to be 20%
4. Expected proportion to be 0.17
5. Least detectable error to be 0.35 Substituting the values, n = 2 (2.8)2 [0.1411] (0.35)2

n = 18.06

To determine the difference in prosthetic complications of CAD-CAM fabricated interim prosthesis as compared to denture conversion prosthesis within 85% of the true value with 95% confidence, a sample size of 18 per group was determined (alpha=0.05).

Approximately 18 subjects per group need to be taken in the present study. To cater for 10% drop-outs, the sample size was adjusted to 20 per group.

9. Planned Analyses

Primary outcomes:

The difference in prosthetic complications between the two groups will be compared using Fisher's exact test.

Secondary Analyses

Secondary outcomes:

The difference in implant survival rates will be evaluated using Kaplan-Meier estimation.

The difference in technical complications will be analyzed using Fisher's exact test and Chi-square test.

Inter group comparison (2 groups) will be done using t-test for peri-implant biological parameters (Probing depth, Plaque control record, Bleeding on probing, marginal bone levels).

Patient-reported outcome measures will be analyzed using Chi-Square test.

Interim Analyses The primary endpoint is at 3 months after BL and the analysis of the data collected up to those visits will be done. No Interim Analysis will be done. However, further analyses will be done after collection of 1-year data, 3- and 5-year data in order to monitor the study outcomes over the time.

10. Safety During the entire duration of the study, all adverse events (AEs), serious adverse events (SAEs) are to be collected, fully investigated and documented in source documents and case report forms (CRF). Study duration encompasses the time from when the participant signs the informed consent until the last investigation plan-specific procedure has been completed.

AE/SAE incidents will be collected at the regular study visits. All adverse events will be documented in a timely manner throughout the clinical investigation and reported as specified in ISO 14155 8.2.5 and 9.8.

ELIGIBILITY:
Inclusion Criteria:

Patients should be of minimum 18 years to be included in the study.

* Patient with edentulous maxilla
* Presence of natural teeth or dentures in the mandibular arch
* Presence of adequate primary stability during implant placement.
* Adequate bone volume to place at least 4 implants with regular platform of at least 6 mm in length
* Presence of at least 6mm (height) of bone in the distal most prosthetic position (in the region of 2nd premolar or 1st molar)
* Presence of at least 8 mm (height) and 6 mm (width) of bone in the anterior region (canine or lateral incisor) to place an implant of a regular diameter and a minimum length of 8 mm.
* Presence of healed maxillary edentulous ridge (at least 3 months post extraction)
* Written informed consent

Exclusion Criteria:

* Self reported history of bruxism
* Uncontrolled diabetes (HbA1c>7.5 mg/dl)
* History of irradiation in the head and neck region
* Inability to comply with annual implant maintenance follow up
* Ridge profile not allowing the placement of a fixed prostheses.
* Presence of any uncontrolled systemic disease that contraindicates implant placement.
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Complications of CAD-CAM prosthesis | 3 months of function
  The primary outcome of the study is the evaluation of prosthetic complications of CAD-CAM fabricated and denture-conversion prosthesis using modified USPHS scores at 3 months of function. USPHS (United States Public Health Service) criteria A, B, C D are used where when rated A an excellent restoration is achieved and D is rated as failure.

SECONDARY OUTCOMES:
Survival rates | 1 year, 3 years and 5 years after insertion of final prosthesis
  To evaluate implant survival rates between group axial and group tilted
Technical outcomes and complications: Prosthetic level | 4 weeks - after insertion of provisional prosthesis; 4 weeks, 1 year, 3 and 5 years after final prosthesis
  They will be evaluated at 4 weeks after insertion of the provisional prosthesis; at 4 weeks, 1 year, 3 years and 5 years after insertion of final prosthesis by using the modified USPHS (United States Public Health Service) criteria. The scale A, B, C D is used where when rated A an excellent restoration is achieved and D is rated as failure.
Technical outcomes and complications: Implant level | 4 weeks - after insertion of provisional prosthesis; 4 weeks, 1 year, 3 and 5 years after final prosthesis
  - Fracture of screw and implant will be evaluated at 4 weeks and 3 months after insertion of provisional prosthesis and at 4 weeks, 1 year, 3 years and 5 years after final prosthesis
VAS provisional prosthesis | 4 weeks - after insertion of provisional prosthesis; 4 weeks, 1 year, 3 and 5 years after final prosthesis
  VAS scores based questionnaires about maintenance of oral hygiene, ability to speak, comfort and aesthetics will be evaluated at 4 weeks after insertion of provisional prosthesis and; after a functional period of 3 months. Visual Analog Scale (VAS) is used with the range from min. 0 up to max. 100, where higher score means better outcome.
Evaluation about ease of surgery | 8 weeks after interim prosthesis insertion
  VAS scores based questionnaires about ease of surgery. Visual Analog Scale (VAS) is used with the range from min. 0 up to max. 100, where higher score means better outcome.
Clinical outcome | 4 weeks and 3 months - after insertion of provisional prosthesis; 4 weeks, 1 year, 3 and 5 years after final prosthesis
  Level of Probing depth (PD, mm)
Radiographic Outcome | 4 weeks and 3 months - after insertion of provisional prosthesis; 4 weeks, 1 year, 3 and 5 years after final prosthesis
  Marginal bone levels (MBL) - the average change in peri-implant bone level will be measured. Peri-apical radiographs will be recorded by using the long-cone paralleling technique and the Rinn XCP extension cone paralleling system (Dentsply Rinn, Elgin, IL, USA).
VAS final prosthesis | 4 weeks - after insertion of provisional prosthesis; 4 weeks, 1 year, 3 and 5 years after final prosthesis
  VAS scores based questionnaires about maintenance of oral hygiene, ability to speak, comfort and aesthetics will be evaluated at 4 weeks after insertion of final prosthesis and; after a functional period of 1, 3 and 5 years. Visual Analog Scale (VAS) is used with the range from min. 0 up to max. 100, where higher score means better outcome.
OHIP-14 final prosthesis | 4 weeks - after insertion of provisional prosthesis; 4 weeks, 1 year, 3 and 5 years after final prosthesis
  OHIP-14 will be evaluated at 4 weeks after insertion of final prosthesis and; after a functional period of 1, 3 and 5 years.
OHIP-14 provisional prosthesis | 4 weeks - after insertion of provisional prosthesis; 4 weeks, 1 year, 3 and 5 years after final prosthesis
  OHIP-14 will be evaluated at 4 weeks after insertion of provisional prosthesis and; after a functional period of 3 months
Evaluation of ease of treatment | 8 weeks after interim prosthesis insertion
  VAS scores based questionnaires about insertion of CAD-CAM fabricated provisional prostheses or denture conversion prostheses will be assessed by the operators after insertion of the implants and insertion of provisional prosthesis. Visual Analog Scale (VAS) is used with the range from min. 0 up to max. 100, where higher score means better outcome.
Clinical outcome | 4 weeks and 3 months - after insertion of provisional prosthesis; 4 weeks, 1 year, 3 and 5 years after final prosthesis
  Rate of Bleeding on probing (BOP, 0/1)
Clinical outcome | 4 weeks and 3 months - after insertion of provisional prosthesis; 4 weeks, 1 year, 3 and 5 years after final prosthesis
  Rate of Plaque control record (PCR, 0/1)

CONTACTS AND LOCATIONS:
Locations (1):
- M.A. Rangoonwala College of Dental Sciences and Research Center, Department of Prosthodontics, Pune, India